CLINICAL TRIAL: NCT00788645
Title: The Use of a Forecasting System for Predicting Exacerbations of COPD: Effect on Symptoms and Hospitalisation and Relevance of Viral Infections
Brief Title: The Use of a Forecasting System for Predicting Exacerbations of COPD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Harsukh Parmar, MD, Early Development Director, RITA, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D6256M00017
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Smoking; COPD; Chronic Obstructive Lung Disease; COPD Exacerbations; Viruses and Bacteria associated with COPD exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Forecast (Experimental): COPD patients receiving advice and poor weather warning
  Interventions: Behavioral: COPD self care advice; Behavioral: Poor weather forecast warning
- No Forecast (Experimental): COPD patients receiving advice and poor weather warning
  Interventions: Behavioral: COPD self care advice
- Control (No Intervention): Age matched non - COPD subjects

INTERVENTIONS:
Behavioral: COPD self care advice — Information leaflets on COPD and thermometers to monitor the ambient temperature in the bedroom and living room
  Arms: Forecast; No Forecast
Behavioral: Poor weather forecast warning — Interactive automated telephone service to contact patients prior to anticipated periods of poor weather
  Arms: Forecast

SUMMARY:
People with Chronic Obstructive Pulmonary Disease (COPD) often have periods during the year when their symptoms become worse. These are often due to an infection and are called "exacerbations" by doctors. Exacerbations are more common in the winter and also seem to be related to particular types of weather. As well as forecasting the weather the UK Met Office has developed a system to try to predict when exacerbations are likely to occur. The main purpose of this research study is to find out whether the Met Office forecasting service can predict when exacerbations are more likely to occur and whether the advice given during the predicted higher risk periods leads to fewer patients having an exacerbation or if it reduces the impact of the exacerbation. The study will also assess if there is a link between viral or bacterial infection and breathing problems that occur during the study period. The study will also collect information about possible causes of the breathing problems and what happens to the person afterwards. The results of this study will help us learn more about breathing problems which may lead to new research studies that would aim to improve the care of people with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smokers with a diagnosis of COPD
* Having impaired lung function as measured by spirometry

Exclusion Criteria:

* History of asthma or nasal symptoms caused by hayfever
* No telephone
* Inability to record symptoms in an electronic diary (PDA)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The incidence and frequency of COPD exacerbations in each of the intervention groups | December 2008 to March 2009 inclusive
Electronic diary symptoms using the EXACT instrument | Daily recording

SECONDARY OUTCOMES:
Medication usage and hospital admissions | Acutely
Changes in the St Georges Respiratory questionaire | Start and end of study period
Severity and duration of exacerbations assessed using the EXACT instrument | Daily recording

CONTACTS AND LOCATIONS:
Overall Officials: David Halpin, MD, Principal Investigator — Royal Devon and Exeter Hospital, Exeter, Devon, UK
Locations (1):
- Research Site, Exeter, United Kingdom

REFERENCES:
- [Derived] Halpin DM, Laing-Morton T, Spedding S, Levy ML, Coyle P, Lewis J, Newbold P, Marno P. A randomised controlled trial of the effect of automated interactive calling combined with a health risk forecast on frequency and severity of exacerbations of COPD assessed clinically and using EXACT PRO. Prim Care Respir J. 2011 Sep;20(3):324-31, 2 p following 331. doi: 10.4104/pcrj.2011.00057. PMID 21687919